## **Statistical Analysis Plan (SAP)**

Official Title: The Effect of Tele-Nursing Service on Patients' Pain and Activity Level in

Patients Diagnosed With Fibromyalgia

Unique Protocol ID: NTK

NCT Number: [NCTXXXXXXXX]

Document Date: August 18, 2025

Sponsor: Çankırı Karatekin University

Principal Investigator: Assist. Prof. Nedret Tekin Kaya

IRB Approval: Çankırı Karatekin University Scientific Research Ethics Committee, Approval

No: 2023/09

Facility Location: Çankırı Karatekin University, Kırkevler Mahallesi, Kastamonu Caddesi,

No:244 Uluyazı Kampüsü 18200 Merkez Çankırı, Turkey

## Statistical analysis

The data were analyzed using IBM SPSS Statistics version 26.0. Group comparisons were performed using independent-samples t-tests and ANOVA. Statistical significance was set at p<0.05. The data were analyzed using IBM SPSS Statistics version 26.0. Group comparisons were performed using independent-samples t-tests and ANOVA. Statistical significance was set at p<0.05. Descriptive data were shown with mean, standard deviation, median, number and percentage. Socio-demographic differences between the intervention and control groups were analyzed using Chi-squared tests for nominal variables and independent samples t-tests for continuous variables. Paired t test was used to determine the difference between two normally distributed groups and independent t test was used for nonnormally distributed variables.